CLINICAL TRIAL: NCT05172869
Title: Comparison of Two Different Approaches in the Fascia Iliaca Compartment Block in Femoral Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Damla kocak, Research Assistant, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Ankara City Hospital
Record Dates: First submitted 2021-10-16; First posted 2021-12-29 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Femoral Fractures; Postoperative Pain
Keywords: Nerve Block [E03.155.086.711]; Femoral Fractures [C26.558.276]; Hip Fractures [C26.558.276.425]; Analgesia [E03.091]; Analgesia, Patient-Controlled [E03.091.120]; Pain, Postoperative [C23.888.592.612.832]; Pain, Procedural [C23.888.592.612.860]; Suprainguinal Fascia Iliaca Block; Infrainguinal Fascia Iliaca Block; Opioid Consumption
MeSH Terms: conditions — Femoral Fractures; Pain, Postoperative; Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: Patients who will undergo surgery will be divided into two randomized groups, each containing 34 patients, in the preoperative unit with a randomization program, as the group in which FICB was applied with the suprainguinal approach (Group S) and the group in which FICB was applied with the infrainguinal approach (Group I).
  FICB can be applied with ultrasound-guided suprainguinal or infrainguinal approaches. Studies on the superiority of the two methods used in clinical practice are limited. In this study, it is aimed to compare the suprainguinal (Group S) and infrainguinal (Group I) approaches of FICB applied in the preoperative period in femoral fractures. These two methods will be compared in terms of postoperative pain scores (11-point numeric scale), morphine consumption (by intravenous patient controlled analgesia for postoperative 24 hours) and possible side effects-complications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S: Suprainguinal Performed FICB (Active Comparator): Suprainguinal Performed FICB
  Interventions: Procedure: Suprainguinal Performed FICB
- Group I: Infrainguinal Performed FICB (Active Comparator): Infrainguinal Performed FICB
  Interventions: Procedure: Infrainguinal Performed FICB

INTERVENTIONS:
Procedure: Suprainguinal Performed FICB — Linear ultrasound probe places above inguinal ligament sagittally, close to the femoral crease and superior-lateral to the femoral artery. It is aimed to spreading local anesthetics under the fascia iliaca medial-laterally
  Arms: Group S: Suprainguinal Performed FICB
Procedure: Infrainguinal Performed FICB — Linear ultrasound probe places below inguinal ligament transversally, close to the femoral crease and lateral to the femoral artery. It is aimed to spreading local anesthetics under the fascia iliaca medial-laterally
  Arms: Group I: Infrainguinal Performed FICB

SUMMARY:
Fascia Iliaca Compartment Block (FICB) is a popular regional anaesthetic technique for surgical procedures involving the hip joint and femur. The FICB may be thought of as an anterior approach to the lumbar plexus where local anaesthetic is injected proximally beneath the fascia iliaca, with the aim of blocking the femoral nerve ,obturator nerve and lateral cutaneous nerve of thigh simultaneously.

In addition to providing effective analgesia, peripheral nerve blocks are increasingly preferred especially in frail patient groups such as the geriatric population which femoral fractures are the most common, because of their advantages such as avoiding the complications of neuraxial anesthesia and the side effects of opioids.

FICB can be applied with ultrasound-guided suprainguinal or infrainguinal approaches. Studies on the superiority of the two methods used in clinical practice are limited. In this study, it is aimed to compare the suprainguinal (Group S) and infrainguinal (Group I) approaches of FICB applied in the preoperative period in femoral fractures in which spinal anesthesia method was chosen. These two methods will be compared in terms of postoperative pain scores (11-point numeric scale), morphine consumption (by intravenous patient controlled analgesia for postoperative 24 hours) and possible side effects-complications.

DETAILED DESCRIPTION:
After ethical committee approval, at least 68 patients who will undergo surgery for femoral fracture will be included in the study. Our study was planned as prospective, randomized, double-blind.

At least 68 patients of both sexes, 18 years of age and older, American Society of Anesthesiologists Score-1,2,3 ( ASA 1,2,3) who will undergo surgery for femoral fracture will be included.

Patients who will undergo surgery will be divided into two randomized groups, each containing 34 patients, in the preoperative unit with a randomization program, as the group in which FICB was applied with the suprainguinal approach (Group S) and the group in which FICB was applied with the infrainguinal approach (Group I).

Routine monitoring [electrocardiogram (ECG), noninNRSive blood pressure, peripheral oxygen saturation (SpO2) measured by pulse oximetry] will be performed for both groups, and heart rate (beats/minute), blood pressure (mmHg), SpO2 (%) will be recorded. Pain intensity, as measured by the 11-Point Numerical Rating Scale (NRS) for pain (0: no pain, 10: worst pain imaginable) will be recorded. All patients in both groups will be administered a mixture of 200mg 2% lidocaine and 0.25% 75mg bupivacaine, with a total volume of 40 ml, with an 80 mm peripheral block needle, accompanied by ultrasonography (US). To avoid toxic doses of local anesthetics, patients with a body weight of less than 50 kg will not be included in the study.

Patients in both groups will undergo sensory examination every 5 minutes for 30 minutes after FICB is performed (sensory: 0, hypoesthesia: 1, no sensation: 2). Sensory examination scoring will be performed and recorded separately for femoral nerve, lateral femoral cutaneous nerve and obturator nerve derivations. Patients with NRS 0-4 and a total sensory scale score for three leads 3 out of 6 will be considered suitable for positioning spinal anesthesia. Among these patients, patients with a sensory scale of 5 and 6 points will be considered as complete block, and their full block duration will be recorded.

The patient will be placed on the operating table in the lateral decubitus position with the fractured side down, and the dynamic NRS (pain score during the lateral decubitus positioning movement with the patient's fractured side down) and static NRS value will be recorded to determine the pain caused by this position. In patients with unsuccessful sensory block application (sensory scale total is 2 or less out of 6, NRS is 5 and above), 0.03 mg/kg midazolam and 1 μg/kg fentanyl will be administered as an intravenous (iv) bolus, and this information will be recorded.

The comfort of the anesthesiologist performing the spinal anesthesia will be recorded (Poor: 0, fair: 1, good: 2, very good: 3).

The heart rate, blood pressure, SpO2 values and pain scores of the patients in both groups will be recorded as static NRS (pain score at rest) before FICB, static NRS and dynamic NRS during position for spinal anesthesia after FICB, and static NRS at the 5th minute after spinal anesthesia.

Heart rate, blood pressure and SpO2 values will be recorded every 15 minutes throughout the operation.

At the end of the operation, the patients will be followed in Postanesthesia Caring Unit (PACU) for the first 24 hours postoperatively. At the end of 24 hours, patients with a Modified Aldrete Score of 9 and above will be transferred to the ward and the follow-up will be terminated.

All patients in both groups will receive intravenous patient-controlled analgesia (PCA) prepared with morphine at the end of the operation. In the PCA device, only the bolus dose program will be selected and it will be prepared with morphine at a concentration of 0.2 mg/ml (30 mg of morphine will be supplemented with 0.09% isotonic saline, so that the total volume will be 150 ml). It will be adjusted as the bolus dose 1 mg, the lock time 20 minutes, the 4-hour limit 8 mg. Basal infusion will not be administered, and when the patient has pain with a NRS score of 5 or more in the postoperative period, bolus administration will be performed with the patient button of the PCA device and each bolus will be recorded by the device. The use of the PCA device will be explained in detail to the patients. Patients whose have pain of NRS 5 and above, but cannot cooperate to press the bolus button (patients who show partial cooperation due to dementia, etc.) a bolus dose will be administered by PACU nurse or anesthesiologist.

Patients will be followed for the first 24 hours with vitals, postoperative pain scores (NRS) and possible opioid side effects related to IV morphine PCA administration. Static and dynamic NRS scores of the patients at 0, 2, 8, 16 and 24 hours postoperatively, at which hour in the postoperative period the first analgesic requirement (time to administer the first bolus dose with the PCA device due to NRS 5 and above), the total amount of opioid consumed during the 24 hours (mg morphine /24 hours) and any side effects (itching, nausea, vomiting, urinary retention, delirium, somnolence, respiratory distress-hypoxia, etc.) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Undergo femoral fracture surgery
* ASA 1-2-3
* 18 years and older
* Accepting preoperative fascia iliaca compartment block application

Exclusion Criteria:

* Patients younger than 18 years
* Patients with an ASA score of 4 and greater than 4
* Patients who are unable to read, understand and sign the consent form
* Patients who do not want to sign the consent form
* Patients deemed unsuitable by the investigator
* Patients with body weight less than 50 kg
* Patients with hypersensitivity to local anesthetics
* Patients with known neuropsychiatric disease
* Patients with coagulopathic disease or anticoagulant drug use that interferes with the application of neuraxial anesthesia or peripheral nerve blockade
* Patients with infection or active skin lesion at the application site of neuraxial anesthesia or peripheral nerve blockade
* Patients who need to be switched to general anesthesia due to spinal anesthesia insufficiency or complications before the operation is completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
Morphine Consumption | 24 hours
  postoperative morphine consumption will be recorded as milligrams for first 24 hours by intravenous patient controlled analgesia (PCA) (mg/24 hours)

SECONDARY OUTCOMES:
Baseline Pain | 0. hours
  11-Point Numerical Rating Scale (NRS) for pain (0: no pain, 10: worst pain imaginable) will be evaluated before applying block
Positional Pain | 0. hours
  After Fascia Iliaca Compartment Block performed, the pain score during the lateral decubitus positioning movement with the patient's fractured side down for performing spinal anesthesia will be recorded by NRS (11-Point Numerical Rating Scale)
Postoperative 2nd Hour Pain | 2. hours
  11-Point Numerical Rating Scale (NRS) for pain (0: no pain, 10: worst pain imaginable) will be evaluated postoperative 2nd hour
Postoperative 8th Hour Pain | 8. hours
  11-Point Numerical Rating Scale (NRS) for pain (0: no pain, 10: worst pain imaginable) will be evaluated postoperative 8th hour
Postoperative 16th Hour Pain | 16. hours
  11-Point Numerical Rating Scale (NRS) for pain (0: no pain, 10: worst pain imaginable) will be evaluated postoperative 16th hour
Postoperative 24th Hour Pain | 24. hours
  11-Point Numerical Rating Scale (NRS) for pain (0: no pain, 10: worst pain imaginable) will be evaluated postoperative 24th hour

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Lafçı, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No